CLINICAL TRIAL: NCT04326023
Title: Myelodysplastic Syndrome and Acute Myeloid Leukemia Related to PARP Inhibitors in Cancer Patients : an Observational and Retrospective Study Using the WHO and the French Pharmacovigilance Databases (MyeloRIB)
Brief Title: Myelodysplastic Syndrome and Acute Myeloid Leukemia Related to PARP Inhibitors (MyeloRIB)
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 20200317
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: PARP Inhibitors — olaparib, rucaparib, niraparib, talazoparib, veliparib

SUMMARY:
Although PARP inhibitors (PARPi) have proved effective in treating many cancers, few patients receiving PARPi may experience rare but life-threatening adverse events such as myelodysplastic syndrome (MDS) and/or acute myeloid leukaemia (AML). Today, data about MDS/AML are scarce.

The objective was to investigate reports of MDS/AML adverse events related to PARPi, including olaparib, rucaparib, niraparib, talazoparib and veliparib using the World Health Organization (WHO) and the French pharmacovigilance databases.

DETAILED DESCRIPTION:
Here, investigators use the World Health Organization (WHO) and the French database of individual safety case reports, to identify cases of MDS/AML related to PARPi.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO, also called VigiBase) or French database of individual safety case reports at the time of the extraction,
* Patients treated with at least 1 PARPi (with ATC classification system): olaparib (ATC L01XX46), niraparib (ATC L01XX54), rucaparib (ATC L01XX55), talazoparib (ATC L01XX60), veliparib (none).

Exclusion Criteria:

* Chronology not compatible between the PARPi and adverse event (MDS/AML)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients treated with PARPi and experiencing MDS/AML.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
MDS/AML reports related to PARPi (from WHO database). | From inception to May 3, 2020
  Identification of the MDS and/or AML adverse event related to PARP inhibitors reported in the World Health Organization (WHO) database of individual safety case reports.
MDS/AML reports related to PARPi (from French database). | From inception to May 1, 2021
  Identification of the MDS and/or AML adverse event related to PARP inhibitors reported in the French pharmacovigilance database of individual safety case reports. The aim is to describe clinical features of these rare adverse events, including bone marrow analyzes, cytogenetic and molecular abnormalities, blasts immunophenotyping anonymously reported in this database.

SECONDARY OUTCOMES:
Description of the median time to onset since first PARPi exposure. | From inception to May 3, 2020
Description of the fatality rate. | From inception to May 3, 2020
Description of patients who experienced co-reported adverse events. | From inception to May 3, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

REFERENCES:
- [Derived] Morice PM, Leary A, Dolladille C, Chretien B, Poulain L, Gonzalez-Martin A, Moore K, O'Reilly EM, Ray-Coquard I, Alexandre J. Myelodysplastic syndrome and acute myeloid leukaemia in patients treated with PARP inhibitors: a safety meta-analysis of randomised controlled trials and a retrospective study of the WHO pharmacovigilance database. Lancet Haematol. 2021 Feb;8(2):e122-e134. doi: 10.1016/S2352-3026(20)30360-4. Epub 2020 Dec 18. PMID 33347814